CLINICAL TRIAL: NCT00626236
Title: A Randomized, Multicenter, Parallel Group, Dose-Ranging Study to Evaluate the Safety and Tolerability of SPN-810 in Children With Attention-Deficit/Hyperactivity Disorder (ADHD) and Persistent Serious Conduct Problems
Brief Title: Phase 2a Study of Safety and Tolerability of SPN-810 in Children With ADHD and Persistent Serious Conduct Problems
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 810P201
Record Dates: First submitted 2008-02-20; First posted 2008-02-29 (Estimated); Results first posted 2025-09-16 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-08

CONDITIONS: Attention Deficit Disorder With Hyperactivity; Conduct Disorder
Keywords: ADHD and conduct problems
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Conduct Disorder | interventions — Molindone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment 1 (Experimental): Treatment 1: SPN-810 5mg/day for subjects <30kg and 10mg/day for subjects ≥30kg
  Interventions: Drug: SPN-810
- Treatment 2 (Experimental): Treatment 2: SPN-810 10mg/day for subjects <30kg and 20mg/day for subjects ≥30kg.
  Interventions: Drug: SPN-810
- Treatment 3 (Experimental): Treatment 3: SPN-810 15mg/day for subjects <30kg and 30mg/day for subjects ≥30kg.
  Interventions: Drug: SPN-810
- Treatment 4 (Experimental): Treatment 4: SPN-810 20mg/day for subjects <30kg and 40mg/day for subjects ≥30kg.
  Interventions: Drug: SPN-810

INTERVENTIONS:
Drug: SPN-810 — 1.67mg capsule taken TID
  Other Names: molindone
  Arms: Treatment 1
Drug: SPN-810 — 3.33mg capsule taken TID
  Other Names: molindone
  Arms: Treatment 2
Drug: SPN-810 — 5mg capsule taken TID
  Other Names: molindone
  Arms: Treatment 3
Drug: SPN-810 — 6.67 mg capsule taken TID
  Other Names: molindone
  Arms: Treatment 4

SUMMARY:
The primary objective was to evaluate the safety and tolerability of four doses of SPN-810 in children with ADHD and persistent serious conduct problems.

DETAILED DESCRIPTION:
This will be a randomized, multicenter, parallel group, dose-ranging safety and tolerability study in children with ADHD and persistent serious conduct problems. The target subjects are healthy male or female children aged 6 to 12 years, inclusive, with a diagnosis of ADHD with persistent serious conduct problems. To determine eligibility for the study, subjects will undergo an initial screening visit. Seventy-two subjects will be randomized in the study; assuming a 17% dropout rate, it is anticipated that 60 subjects will complete the study. The study will consist of a Screening Period (within 28 days prior to the first dose administration), a Titration Period of 2 to 5 weeks, a Maintenance Period of 6 weeks, and a Safety Follow-up, which will be performed 30 days after the final study visit. The total subject duration in the study will be 16 to 19 weeks depending on the treatment group assignment. The total study duration is anticipated to be 15.5 months. A total of 72 subjects will be randomized based on weight at baseline, to 1 of 4 treatment groups.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy pediatric male or female subjects, age 6 to 12 years.
2. Diagnostic and Statistical Manual of Mental Disorders - IV -Text Revision (DSM-IV-TR) diagnosis of ADHD.
3. NCBRF-TIQ disruptive behavior disorder subscale 27 or greater at baseline; AND a score of 2 or more on at least 1 of the following 3 items of the conduct problem subscale: knowingly destroys property, gets in physical fights, physically attacks people.
4. IQ greater than 71.

Exclusion Criteria:

1. Current or lifetime diagnosis of bipolar disorder, post-traumatic stress disorder, personality disorder, or psychosis not otherwise specified.
2. Currently meeting DSM-IV-TR criteria for major depressive disorder, obsessive compulsive disorder, or pervasive developmental disorder.
3. Any other anxiety disorder as primary diagnosis.
4. Use of anticonvulsants, antidepressants, lithium, carbamazepine, valproic acid, or cholinesterase inhibitors within 2 weeks of baseline.
5. Unstable endocrinological or neurological conditions which confound the diagnosis or are a contraindication to treatment with antipsychotics.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 2008-10-21 (Actual); Primary Completion 2009-09-23 (Actual); Study Completion 2009-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Findling, MD, Principal Investigator — University Hospitals Case Medical Center/Case Western Reserve University
Locations (9):
- United States (9):
  - Florida Clinical Research Center, Bradenton, Florida
  - Sarkis Clinical Trials, Gainesville, Florida
  - CNS Healthcare, Orlando, Florida
  - Capstone Clinical Research, Libertyville, Illinois
  - The Psychopharm Research Cntr - LSU Dept of Psychiatry, Shreveport, Louisiana
  - IPS Research, Oklahoma City, Oklahoma
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - Alliance Research Group, Richmond, Virginia
  - Northwest Clinical Trials, Bellevue, Washington

REFERENCES:
- [Derived] Stocks JD, Taneja BK, Baroldi P, Findling RL. A phase 2a randomized, parallel group, dose-ranging study of molindone in children with attention-deficit/hyperactivity disorder and persistent, serious conduct problems. J Child Adolesc Psychopharmacol. 2012 Apr;22(2):102-11. doi: 10.1089/cap.2011.0087. Epub 2012 Feb 28. PMID 22372512
- See also: A phase 2a randomized, parallel group, dose-ranging study of molindone in children with attention-deficit/hyperactivity disorder and persistent, serious conduct problems — https://pubmed.ncbi.nlm.nih.gov/22372512/

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment 1 5/10mg TDD: SPN-810: capsule taken three times a day
- Treatment 2 10/20mg TDD; Treatment 3 15/30mg TDD; Treatment 4 20/40mg TDD: SPN-810: capsule taken TID
Period: Overall Study
Arm/Group | Treatment 1 5/10mg TDD | Treatment 2 10/20mg TDD | Treatment 3 15/30mg TDD | Treatment 4 20/40mg TDD
Started | 20 | 19 | 19 | 20
Completed | 14 | 12 | 15 | 14
Not Completed | 6 | 7 | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment 1 5/10mg TDD | Treatment 2 10/20mg TDD | Treatment 3 15/30mg TDD | Treatment 4 20/40mg TDD | Total
Number analyzed (Participants) | 20 | 19 | 19 | 20 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.5 (1.88) | 9.4 (1.98) | 8.8 (2.12) | 8.8 (2.00) | 8.8 (1.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 6 | 1 | 11
  Male | 19 | 16 | 13 | 19 | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 5 | 1 | 7
  Not Hispanic or Latino | 19 | 19 | 14 | 19 | 71
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 9 | 8 | 9 | 7 | 33
  White | 11 | 11 | 8 | 13 | 43
  More than one race | 0 | 0 | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 19 | 19 | 20 | 78

OUTCOME MEASURES:

1. Primary Outcome: The Nisonger Child Behavior Rating Form- Typical Intelligence Quotient (NCBRF-TIQ) Conduct Problem Subscale Score
Description: The Nisonger Child Behavior Rating Form (NCBRF) is an instrument designed to assess the behavior of children with intellectual or developmental disabilities. The NCBRF-TIQ is a 66-item behavior rating form designed to assess the behavior of children and adolescents with typical development. The NCBRF is made up of three sections: I, Where raters can identify unusual circumstances that may have affected the youth's behavior; II, where positive behaviors are rated, and III, a listing of problem behaviors. There are separate Teacher and Parent versions of the form, and the NCBRF takes about 15 minutes to complete. The NCBRF is designed to be used with children and adolescents ages 3 to 16 years. The lowest score is a "0" and the highest score is "198". A higher score of the Conduct Problem Subscale score means a worse outcome. A change or negative score means improvement. Data represent the change from baseline (Visit 1) and 11 time points (Visit 2 to Visit 12).
Time Frame: Weekly visits starting from Visit 1 (Week 1) to Visit 12 (12 weeks)
Population: ITT population consisted of all Safety Population subjects with at least 1 post-baseline efficacy assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment 1 5/10mg TDD | Treatment 2 10/20mg TDD | Treatment 3 15/30mg TDD | Treatment 4 20/40mg TDD
Number analyzed (Participants) | 20 | 19 | 19 | 20
score on a scale
  Mean Score at Baseline | 20.4 (5.22) | 25.7 (6.98) | 26.0 (5.51) | 26.0 (7.63)
  Visit 2 Change from Baseline | -0.6 (5.82) | -3.3 (5.94) | -2.6 (6.69) | -3.3 (5.72)
  Visit 3 Change from Baseline | -0.6 (5.82) | -7.1 (9.95) | -3.4 (6.78) | -6.1 (6.69)
  Visit 4 Change from Baseline | -0.6 (5.82) | -7.1 (9.95) | -5.0 (9.57) | -8.9 (6.95)
  Visit 5 Change from Baseline | -0.6 (5.82) | -7.1 (9.95) | -5.0 (9.57) | -11.7 (7.68)
  Visit 6 Change from Baseline | -2.7 (5.38) | -7.8 (9.60) | -6.4 (9.31) | -11.6 (7.51)
  Visit 7 Change from Baseline | -4.8 (6.07) | -8.1 (9.79) | -7.6 (8.71) | -12.9 (8.35)
  Visit 8 Change from Baseline | -6.0 (7.19) | -7.6 (8.37) | -9.0 (9.84) | -14.5 (9.24)
  Visit 9 Change from Baseline | -8.1 (6.33) | -7.8 (8.21) | -9.7 (9.74) | -14.8 (8.49)
  Visit 10 Change from Baseline | -7.9 (6.86) | -7.9 (8.36) | -11.2 (8.93) | -13.6 (9.87)
  Visit 11 Change from Baseline | -7.9 (6.77) | -9.9 (9.31) | -9.2 (10.60) | -14.5 (8.65)
  Visit 12 Change from Baseline | -7.0 (7.13) | -8.7 (9.31) | -8.2 (10.51) | -14.3 (8.64)

2. Secondary Outcome: The Changes From Baseline in the CGI-S
Description: The CGI scale was developed to provide a brief, stand-alone assessment of the clinician's view of a subject's global functioning prior to and after the administration of study medication. The severity of illness (CGI-S) is rated by the investigator on a 7-point scale with 1=Normal, 2=Borderline ill, 3=Mildly ill, 4=Moderately ill, 5=Markedly ill, 6=Severely ill, and 7=Extremely ill. Data represent the change from baseline (Visit 1) and 11 time points (Visit 2 to Visit 12). A lower overall score in subsequent testing indicates successful therapy.
Time Frame: Weekly visits starting from Visit 1 (Week 1) to Visit 12 (12 weeks)
Population: ITT population consisted of all Safety Population subjects with at least 1 post-baseline efficacy assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment 1 5/10mg TDD | Treatment 2 10/20mg TDD | Treatment 3 15/30mg TDD | Treatment 4 20/40mg TDD
Number analyzed (Participants) | 20 | 19 | 19 | 20
score on a scale
  Baseline Score | 4.35 (0.587) | 4.74 (0.562) | 4.63 (0.684) | 4.70 (0.470)
  Visit 2 Change From Baseline | -0.20 (0.523) | -0.26 (0.562) | -0.11 (0.459) | -0.20 (0.523)
  Visit 3 Change From Baseline | -0.20 (0.523) | -0.47 (0.772) | -0.37 (0.496) | -0.45 (0.510)
  Visit 4 Change From Baseline | -0.20 (0.523) | -0.47 (0.772) | -0.63 (0.831) | -0.75 (0.716)
  Visit 5 Change From Baseline | -0.20 (0.523) | -0.47 (0.772) | -0.63 (0.831) | -1.10 (0.788)
  Visit 6 Change From Baseline | -0.20 (0.523) | -0.68 (0.749) | -0.89 (0.809) | -1.30 (0.923)
  Visit 7 Change From Baseline | -0.55 (0.686) | -0.79 (0.713) | -1.26 (0.991) | -1.30 (0.923)
  Visit 8 Change From Baseline | -0.85 (0.813) | -0.79 (0.855) | -1.37 (0.895) | -1.50 (1.192)
  Visit 9 Change From Baseline | -1.05 (0.759) | -0.89 (0.875) | -1.32 (0.946) | -1.70 (1.218)
  Visit 10 Change From Baseline | -1.10 (0.968) | -0.84 (0.898) | -1.53 (0.964) | -1.65 (1.137)
  Visit 11 Change From Baseline | -1.15 (0.875) | -1.05 (0.970) | -1.37 (1.012) | -1.55 (1.099)
  Visit 12 Change From Baseline | -1.00 (0.973) | -1.00 (1.000) | -1.26 (0.933) | -1.75 (1.293)

3. Secondary Outcome: Clinical Global Impression - Improvement Scale (CGI-I)
Description: Clinical Global Impression Scale. CGI-I is measured relative to the condition at the Baseline on a 7-point scale with 1=Very much improved, 2=Much improved, 3=Minimally improved, 4=No change, 5=Minimally worse, 6=Much worse, and 7=Very much worse. A lower overall score in subsequential testing indicates successful treatment. Data represent the change from baseline (Visit 1) and 11 time points (Visit 2 to Visit 12).
Time Frame: Weekly visits starting from Visit 1 (Week 1) to Visit 12 (12 weeks)
Population: ITT population consisted of all Safety Population subjects with at least 1 post-baseline efficacy assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment 1 5/10mg TDD | Treatment 2 10/20mg TDD | Treatment 3 15/30mg TDD | Treatment 4 20/40mg TDD
Number analyzed (Participants) | 20 | 19 | 19 | 20
score on a scale
  Visit 2 Change from Baseline | 0.00 (0.0) | 0.00 (0.0) | 0.00 (0.0) | 0.00 (0.0)
  Visit 3 Change from Baseline | 0.00 (0.000) | -0.41 (0.795) | -0.21 (0.631) | -0.42 (0.961)
  Visit 4 Change from Baseline | 0.00 (0.000) | -0.41 (0.795) | -0.58 (0.961) | -0.68 (0.820)
  Visit 5 Change from Baseline | 0.00 (0.000) | -0.41 (0.795) | -0.58 (0.961) | -1.16 (1.167)
  Visit 6 Change from Baseline | -0.12 (0.697) | -0.76 (0.903) | -0.79 (0.918) | -1.26 (1.046)
  Visit 7 Change from Baseline | -0.59 (0.939) | -0.88 (1.111) | -1.21 (0.918) | -1.26 (1.046)
  Visit 8 Change from Baseline | -0.88 (0.928) | -0.88 (1.219) | -1.42 (1.017) | -1.26 (1.098)
  Visit 9 Change from Baseline | -1.06 (0.827) | -0.94 (1.144) | -1.26 (0.933) | -1.37 (1.012)
  Visit 10 Change from Baseline | -1.00 (1.118) | -0.88 (1.317) | -1.53 (1.073) | -1.42 (1.017)
  Visit 11 Change from Baseline | -1.29 (0.985) | -0.94 (1.435) | -1.32 (1.003) | -1.37 (1.012)
  Visit 12 Change from Baseline | -1.12 (1.219) | -1.00 (1.000) | -1.26 (0.872) | -1.32 (1.057)

4. Secondary Outcome: SNAP-IV ADHD Inattention
Description: The ratings from the SNAP-IV scale are grouped into the following 3 subscales: ADHD-Inattention (items #1-9), ADHD-Hyperactivity/Impulsivity (items #10-18), and ADHD combined (items #0-18) Subscales. The symptoms are scored on a 4-point scale. Each subscale score is the average rating of the items scores for the subscale. For the inattention subscale, the scores range from 0-27, the higher the score, the worse the outcome.
  A decrease in score means improvement. Data represent the change between Baseline (Visit 1) to Visit 2, Visit 4, Visit 6, Visit 10 and Visit 12.
Time Frame: Weekly visits starting from Visit 1 (Week 1) to Visit 12 (12 weeks)
Population: ITT population consisted of all Safety Population subjects with at least 1 post-baseline efficacy assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment 1 5/10mg TDD | Treatment 2 10/20mg TDD | Treatment 3 15/30mg TDD | Treatment 4 20/40mg TDD
Number analyzed (Participants) | 20 | 19 | 19 | 20
score on a scale
  Baseline Score | 18.20 (6.810) | 20.42 (4.501) | 20.00 (4.190) | 21.05 (4.211)
  Visit 2 Change from Baseline | -1.55 (5.010) | -1.74 (4.593) | -1.84 (5.167) | 0.10 (5.200)
  Visit 3 Change from Baseline | -1.55 (5.010) | -3.79 (5.149) | -3.84 (4.729) | -1.35 (5.234)
  Visit 4 Change from Baseline | -1.55 (5.010) | -3.79 (5.149) | -5.11 (5.517) | -2.35 (5.770)
  Visit 5 Change from Baseline | -1.55 (5.010) | -3.79 (5.149) | -5.11 (5.517) | -5.30 (7.420)
  Visit 6 Change from Baseline | -1.15 (5.556) | -4.21 (5.583) | -7.16 (4.752) | -5.60 (5.888)
  Visit 7 Change from Baseline | -2.55 (5.104) | -5.84 (4.729) | -6.42 (5.984) | -6.00 (7.732)
  Visit 8 Change from Baseline | -3.95 (6.126) | -5.68 (5.197) | -7.05 (6.302) | -6.65 (7.088)
  Visit 9 Change from Baseline | -5.65 (6.385) | -4.42 (4.706) | -7.05 (5.902) | -8.30 (7.794)
  Visit 10 Change from Baseline | -5.15 (7.206) | -5.42 (4.834) | -8.89 (6.341) | -7.55 (8.733)
  Visit 11 Change from Baseline | -5.65 (7.006) | -5.63 (5.058) | -8.11 (6.420) | -8.20 (7.885)
  Visit 12 Change from Baseline | -4.35 (6.150) | -6.32 (5.558) | -6.84 (5.956) | -8.15 (7.611)

5. Secondary Outcome: SNAP-IV Subscales ADHD Hyperactivity/Impulsivity
Description: The ratings from the SNAP-IV scale are grouped into the following 3 subscales: ADHD-Inattention (items #1-9), ADHD-Hyperactivity/Impulsivity (items #10-18), and ADHD combined (items #1-18) Subscales. The symptoms are scored on a 4-point scale. Each subscale score is the average rating of the items scores for the subscale. For the Hyperactivity/Impulsivity subscale, the scores range from 0-27, the higher the score, the worse the outcome.
  A decrease in score means improvement. Data represent the change between Baseline (Visit 1) to Visit 2, Visit 4, Visit 6, Visit 10 and Visit 12.
Time Frame: Weekly visits starting from Visit 1 (Week 1) to Visit 12 (12 weeks)
Population: ITT population consisted of all Safety Population subjects with at least 1 post-baseline efficacy assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment 1 5/10mg TDD | Treatment 2 10/20mg TDD | Treatment 3 15/30mg TDD | Treatment 4 20/40mg TDD
Number analyzed (Participants) | 20 | 19 | 19 | 20
score on a scale
  Baseline Score | 19.60 (5.933) | 21.74 (5.173) | 19.11 (5.517) | 20.95 (4.989)
  Visit 2 Change from Baseline | -0.90 (4.166) | -1.47 (3.821) | -1.42 (4.562) | -1.05 (3.832)
  Visit 3 Change from Baseline | -0.90 (4.166) | -3.32 (4.785) | -3.47 (6.123) | -2.05 (4.915)
  Visit 4 Change from Baseline | -0.90 (4.166) | -3.32 (4.785) | -3.74 (6.814) | -3.80 (5.483)
  Visit 5 Change from Baseline | -0.90 (4.166) | -3.32 (4.785) | -3.74 (6.814) | -5.85 (6.706)
  Visit 6 Change from Baseline | -2.30 (4.802) | -4.16 (5.367) | -5.37 (5.510) | -6.05 (5.520)
  Visit 7 Change from Baseline | -3.90 (4.909) | -4.84 (4.598) | -5.32 (5.991) | -7.10 (7.826)
  Visit 8 Change from Baseline | -5.25 (6.624) | -4.47 (4.439) | -6.21 (6.545) | -7.60 (7.408)
  Visit 9 Change from Baseline | -7.00 (6.383) | -3.79 (4.379) | -5.79 (5.534) | -9.10 (7.594)
  Visit 10 Change from Baseline | -5.90 (6.656) | -5.16 (5.449) | -8.26 (6.393) | -8.35 (7.271)
  Visit 11 Change from Baseline | -6.65 (6.620) | -5.47 (4.846) | -6.37 (6.576) | -9.00 (7.691)
  Visit 12 Change from Baseline | -5.55 (6.739) | -5.79 (5.442) | -5.42 (6.963) | -8.50 (7.309)

6. Secondary Outcome: SNAP-IV Subscales - ADHD Combined
Description: The ratings from the SNAP-IV scale are grouped into the following 3 subscales: ADHD-Inattention (items #1-9), ADHD-Hyperactivity/Impulsivity (items #10-18), and ADHD combined (items #1-18) Subscales. The symptoms are scored on a 4-point scale. Each subscale score is the average rating of the items scores for the subscale. For the combined subscale, the scores range from 0-54, the higher the score, the worse the outcome.
  A decrease in score means improvement. Data represent the change between Baseline (Visit 1) to Visit 2, Visit 4, Visit 6, Visit 10 and Visit 12.
Time Frame: Weekly visits starting from Visit 1 (Week 1) to Visit 12 (12 weeks)
Population: ITT population consisted of all Safety Population subjects with at least 1 post-baseline efficacy assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Treatment 1 5/10mg TDD: SPN-810: capsule taken three times a day (TID)
Arm/Group | Treatment 1 5/10mg TDD | Treatment 2 10/20mg TDD | Treatment 3 15/30mg TDD | Treatment 4 20/40mg TDD
Number analyzed (Participants) | 20 | 19 | 19 | 20
score on a scale
  Baseline Score | 37.80 (11.414) | 42.16 (7.537) | 39.11 (8.888) | 42.00 (8.240)
  Visit 2 Change from Baseline | -2.45 (7.957) | -3.21 (7.627) | -3.26 (8.736) | -0.95 (8.420)
  Visit 3 Change from Baseline | -2.45 (7.957) | -7.11 (9.579) | -7.32 (9.995) | -3.40 (9.338)
  Visit 4 Change from Baseline | -2.45 (7.957) | -7.11 (9.579) | -8.84 (11.758) | -6.15 (10.569)
  Visit 5 Change from Baseline | -2.45 (7.957) | -7.11 (9.579) | -8.84 (11.758) | -11.15 (13.287)
  Visit 6 Change from Baseline | -3.45 (9.854) | -8.37 (10.073) | -12.53 (9.697) | -11.65 (10.554)
  Visit 7 Change from Baseline | -6.45 (9.361) | -10.68 (8.838) | -11.74 (11.293) | -13.10 (15.082)
  Visit 8 Change from Baseline | -9.20 (12.194) | -10.16 (8.902) | -13.26 (12.355) | -14.25 (13.845)
  Visit 9 Change from Baseline | -12.65 (12.006) | -8.21 (8.203) | -12.84 (10.678) | -17.40 (14.702)
  Visit 10 Change from Baseline | -11.05 (13.477) | -10.58 (9.371) | -17.16 (11.701) | -15.90 (15.362)
  Visit 11 Change from Baseline | -12.30 (13.111) | -11.11 (8.730) | -14.47 (12.294) | -17.20 (14.877)
  Visit 12 Change from Baseline | -9.90 (12.251) | -12.11 (9.944) | -12.26 (12.596) | -16.65 (14.203)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from first dose through 7 days after last dose for non-serious AEs, and through 30 days post-treatment for SAEs (total study duration 16-19 weeks including follow-up
Description: All AEs were collected from time of informed consent through 7 days after last dose (non-serious) and through 30-day follow-up (serious AEs). Events were coded using MedDRA Version 11.1.
Arm/Group | Treatment 1 5/10mg TDD | Treatment 2 10/20mg TDD | Treatment 3 15/30mg TDD | Treatment 4 20/40mg TDD
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/19 | 0/19 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19 | 1/19 | 1/20
Other Adverse Events (participants affected / at risk) | 12/20 | 15/19 | 17/19 | 17/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment 1 5/10mg TDD (N=20) | Treatment 2 10/20mg TDD (N=19) | Treatment 3 15/30mg TDD (N=19) | Treatment 4 20/40mg TDD (N=20)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abnormal behavior (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Abnormal behavior was incorrectly recorded as behavioral activation
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment 1 5/10mg TDD (N=20) | Treatment 2 10/20mg TDD (N=19) | Treatment 3 15/30mg TDD (N=19) | Treatment 4 20/40mg TDD (N=20)
Somnolence (Nervous system disorders) | 1 | 1 | 5 | 3
Abdominal pain upper (Gastrointestinal disorders) | 2 | 4 | 1 | 2
Weight decreased (General disorders) | 0 | 2 | 3 | 3
Upper Resipiratory Tract Infection (Reproductive system and breast disorders) | 2 | 1 | 3 | 1
Insomnia (Psychiatric disorders) | 2 | 2 | 1 | 2
Fatigue (General disorders) | 2 | 0 | 1 | 4
Headache (General disorders) | 1 | 0 | 1 | 3
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1 | 2 | 0
Akathisia (Nervous system disorders) | 1 | 0 | 2 | 1
Sedation (Nervous system disorders) | 0 | 0 | 0 | 4
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2
Viral infection (Infections and infestations) | 0 | 2 | 2 | 0
Pyrexia (General disorders) | 0 | 2 | 1 | 1
Pain in extremity (General disorders) | 1 | 0 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Statistical Analysis Plan (2009-08-31): https://cdn.clinicaltrials.gov/large-docs/36/NCT00626236/SAP_000.pdf